CLINICAL TRIAL: NCT03824002
Title: Arterial Stiffness and Endothelial Function Indexes, Relationships With Clinical and Laboratory Variables in a Group of Diabetic Patients in Treatment With Dulaglutide: a Case-control Study
Brief Title: Dulaglutide in Diabetic Patients, Relationship Between Arterial Stiffness, Endothelial Function, Clinical and Laboratory Variables
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, University professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21772
Record Dates: First submitted 2018-12-06; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; dulaglutide; endothelial function
MeSH Terms: conditions — Diabetes Mellitus | interventions — dulaglutide; Insulin Aspart; Insulin Glargine; Metformin; repaglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients treated with dulaglutide (Experimental): Diabetes therapy with dulaglutide and various combinations of aspart insulin, glargine, metformin, repaglinide
  Interventions: Drug: Dulaglutide; Drug: Aspart insulin; Drug: Glargine; Drug: Metformin; Drug: Repaglinide
- patients not treated with dulaglutide (Active Comparator): Diabetes therapy with various combinations of aspart insulin, glargine, metformin, repaglinide but without dulaglutide
  Interventions: Drug: Aspart insulin; Drug: Glargine; Drug: Metformin; Drug: Repaglinide

INTERVENTIONS:
Drug: Dulaglutide — Diabetes therapy with dulaglutide and various combinations of insulin, metformin, glinides
  Other Names: aspart insulin; glargine insulin; metformin; repaglinide
  Arms: patients treated with dulaglutide
Drug: Aspart insulin — Diabetes therapy with various combinations of insulin, metformin, glinides but without dulaglutide
Drug: Glargine — Diabetes therapy with various combinations of insulin, metformin, glinides but without dulaglutide
Drug: Metformin — Diabetes therapy with various combinations of insulin, metformin, glinides but without dulaglutide
Drug: Repaglinide — Diabetes therapy with various combinations of insulin, metformin, glinides but without dulaglutide

SUMMARY:
The study aims to evaluate arterial stiffness and endothelial function indexes and their relationship with clinic and laboratory varible in a group of diabetic patients in treatment with dulaglutide

DETAILED DESCRIPTION:
46 patients with type 2 diabetes mellitus were recruited at the Internal Medicine with Stroke care ward of the University hospital of Palermo "P. Giaccone" from April 2017 to April 2018. For all patients treatment with dulaglutide was undertaken. As control group were recruited 46 patients from the same ward not affected by diabetes mellitus or affected by diabetes mellitus but not in treatment with dulaglutide.

The study was carried out in accordance with the principles of the Helsinki Declaration revised in 2001 and all patients gave their written consent to take part in this research.

Each patient treated with dulaglutide was compared for age, sex and cardiovascular risk with control patients. The diagnosis of type 2 diabetes mellitus was based on the revised criteria of the American Diabetes Association (ADA), and using a clinical algorithm that considered the age of onset of the disease, the symptoms and weight present, the family history and the therapy practiced. Arterial hypertension was defined according to the 2017 ESC-ESH criteria. Dyslipidemia was defined based on total cholesterol levels> 200 mg/dl, triglycerides> 150 mg/dl and HDL levels <40 mg/dl regardless of the patient's gender.

Among the cases enrolled, 46 (100%) had type 2 diabetes mellitus, 37 (80.43%) had arterial hypertension and 26 (56.52%) hypercholesterolemia.

Clinical and anthropometric data were collected at the time of recruitment. Blood samples were taken from each patient (cases and controls) to determine serum glucose, HbA1c, total cholesterol, HDL and LDL cholesterol, triglycerides, creatinine, and a urine sample to assess the presence of microalbuminuria. These withdrawals were then repeated three months and nine months from the time of recruitment.

The digital endothelial function was evaluated through the RHI-pat analysis using Endo-PAT2000. Pulse Wave Velocity (PWV) Carotid-Femoral Pulse was measured in the supine position using an automatic device (SphygmoCor version 7.1) that evaluated the propagation time of the sphygmic wave between the carotid and femoral pulse.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus

Exclusion Criteria:

* cancer, severe ckd, end stage liver disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Reactive Hyperemia Index at 3 and 9 months | 0 months, 3 months and 9 months
  Endothelial function index RHI

SECONDARY OUTCOMES:
Change from Baseline systolic blood pressure at 3 and 9 months | 0 months, 3 months and 9 months
  systolic blood pressure in mmHg
Change from Baseline Body Mass Index at 3 and 9 months | 0 months, 3 months and 9 months
  weight and height will be combined to report BMI in kg/m^2
Change from Baseline cholesterol at 3 and 9 months | 0 months, 3 months and 9 months
  blood cholesterol in mg/dl
Change from Baseline triglycerides at 3 and 9 months | 0 months, 3 months and 9 months
  blood triglycerides in mg/dl
Change from Baseline glucose at 3 and 9 months | 0 months, 3 months and 9 months
  fasting blood glucose in mg/dl
Change from Baseline diastolic blood pressure at 3 and 9 months | 0 months, 3 months and 9 months
  diastolic blood pressure in mmHg
Change from Baseline Pulse Wave Velocity at 3 and 9 months | 0 months, 3 months and 9 months
  Pulse Wave Velocity in m/s

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Ward, University of Palermo, Palermo, Italy

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952